CLINICAL TRIAL: NCT02562482
Title: Phase 2 Randomized, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of a Chikungunya Virus-Like Particle Vaccine, VRC-CHKVLP059-00-VP, in Healthy Adults
Brief Title: Trial for Safety and Immunogenicity of a Chikungunya Vaccine, VRC-CHKVLP059-00-VP, in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VRC 704
Record Dates: First submitted 2015-09-21; First posted 2015-09-29 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Chikungunya Virus Infection
Keywords: Antibody Response; Immune Response; Healthy Volunteer; Vaccine-Mediated Protection; Chikungunya Virus; Vaccines, Virus-like Particles
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: VRC-CHKVLP059-00-VP 20 mcg (Experimental): Group 1 subjects were randomized to receive two intramuscular (IM) injections of CHIKV VLP vaccine (VRC-CHKVLP059-00-VP) at Day 0 and Day 28 (+14 days) at a dose of 20 micrograms (mcg).
  Interventions: Biological: VRC-CHKVLP059-00-VP
- Group 2: Placebo (VRC-PBSPLA043-00-VP) (Placebo Comparator): Group 2 subjects were randomized to receive two intramuscular (IM) injections of Phosphate Buffered Saline (VRC-PBSPLA043-00-VP) placebo at Day 0 and Day 28 (+14 days).
  Interventions: Other: VRC-PBSPLA043-00-VP

INTERVENTIONS:
Biological: VRC-CHKVLP059-00-VP — VRC-CHKVLP059-00-VP is a virus-like particle (VLP) vaccine that consists of CHIKV VLP composed of E1, E2 and capsid proteins of the CHIKV (strain 37997).
  Arms: Group 1: VRC-CHKVLP059-00-VP 20 mcg
Other: VRC-PBSPLA043-00-VP — VRC-PBSPLA043-00-VP, a sterile phosphate buffered saline (PBS) is the placebo for the CHIKV VLP vaccine.
  Arms: Group 2: Placebo (VRC-PBSPLA043-00-VP)

SUMMARY:
This is a multicenter, randomized, placebo-controlled, double-blind study to evaluate the safety and immunogenicity of a 2-injection vaccine Chikungunya virus (CHIKV) virus-like particle vaccine (CHIKV VLP) in healthy adults.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, placebo-controlled, double-blind study to evaluate the safety and immunogenicity of a 2-injection vaccine regimen (Day 0 and 28) with Chikungunya virus (CHIKV) virus-like particle vaccine (CHIKV VLP, VRC-CHKVLP059-00-VP) in healthy adults ages 18-60 years old that reside in CHIKV endemic regions.

The hypothesis is that the vaccine regimen is safe and induces a neutralizing antibody response to CHIKV. The primary objectives are to evaluate safety and tolerability of a 2-injection investigational vaccine regimen of VRC-CHKVLP059-00-VP at 20 mcg compared to placebo (PBS) in healthy adults in CHIKV endemic areas. The secondary objective is to evaluate neutralizing antibody response in vaccine recipients. The exploratory objectives relate to assessing incidence of CHIKV infection in vaccine and placebo recipients, as well as antigen-specific humoral and cellular immune responses during the study.

The expected study duration per subject is approximately 72 weeks with intramuscular (IM) injections scheduled at Day 0 and Day 28.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following criteria:

* 18 to 60 years old
* Available for clinical follow-up through Study Week 72
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
* Able and willing to complete the informed consent process
* Willing to donate blood for sample storage to be used for future research
* In good general health, with a body mass index (BMI)≤40, without clinically significant medical history, and has satisfactorily completed screening
* Physical examination and laboratory results without clinically significant findings within the 56 days prior to enrollment

Laboratory Criteria within 56 days prior to enrollment:

* Hemoglobin either within institutional normal limits or accompanied by site physician approval as consistent with healthy adult status
* White blood cells either within institutional normal range or accompanied by site physician approval as consistent with healthy adult status
* Platelets = 125,000 - 500,000/mm3
* Alanine aminotransferase (ALT) ≤ 1.25 x upper limit of normal (ULN)
* Serum creatinine ≤ 1.1 x ULN based on site institutional normal range
* Negative result on a human immunodeficiency virus (HIV) test that meets local standards for identification of HIV infection
* Negative result on the Chikungunya virus (CHIKV) screening antibody assay.

Criteria applicable to women of childbearing potential:

* Negative human chorionic gonadotropin pregnancy test (urine or serum) on day of enrollment
* Agree to use an effective means of birth control from 21 days prior to enrollment through 12 weeks after the last study injection

Exclusion Criteria:

A subject will be excluded if one or more of the following conditions apply:

Women Specific:

-Planning to become pregnant during the 16 weeks after enrollment in the study

Subject has received any of the following substances:

* Systemic immunosuppressive medications within 2 weeks prior to enrollment
* Blood products within 16 weeks prior to enrollment
* Immunoglobulin within 8 weeks prior to enrollment
* Prior vaccinations with an investigational CHIKV vaccine
* Investigational research agents within 4 weeks prior to enrollment
* Any vaccination within 2 weeks prior to enrollment
* Current anti-tuberculosis (TB) prophylaxis or therapy

Subject has a history of any of the following clinically significant conditions:

* A history of immune-mediated or clinically significant arthritis
* Serious reactions to vaccines that preclude receipt of study injections as determined by the investigator
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
* Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that is expected to require the use of oral or intravenous corticosteroids
* Diabetes mellitus (type I or II), with the exception of gestational diabetes
* Idiopathic urticaria within the past year
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with intramuscular (IM) injections or blood draws
* Malignancy that is active or history of a malignancy that is likely to recur during the period of the study
* Seizure in the past 3 years or treatment for a seizure disorder within the last 3 years
* Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
* Psychiatric condition that may preclude compliance with the protocol; past or present psychoses; or a history of suicide plan or attempt within the five years prior to enrollment
* Any medical or social condition that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rosario, MD, Principal Investigator — San Juan Hospital; Clemente Diaz, MD, Principal Investigator — Puerto Rico Clinical and Translational Research Consortium; Bruno Hoen, MD, Principal Investigator — University Hospital Pointe-a-Pitre, Guadeloupe; Yeycy Donastorg, MD, Principal Investigator — Instituto Dermatológico y Cirugía de Piel; Jean W Pape, MD, Principal Investigator — Centres GHESKIO, Haiti; Andre Cabie, MD, Principal Investigator — Centre Hospitalier Universitaire (CHU), Martinique; Julie Ledgerwood, DO, Study Chair — VRC, NIAID, NIH; Grace Chen, MD, Study Chair — VRC, NIAID, NIH
Locations (6):
- Instituto Dermatológico y Cirugía de Piel, Santo Domingo, Dominican Republic
- University Hospital of Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe
- Centres GHESKIO, Port-au-Prince, Haiti
- Centre Hospitalier Universitaire (CHU), Martinique, Fort-de-France, Martinique
- Puerto Rico (2):
  - San Juan Hospital, Research Unit, Rio Piedras
  - Puerto Rico Clinical and Translational Research Consortium, San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang LJ, Dowd KA, Mendoza FH, Saunders JG, Sitar S, Plummer SH, Yamshchikov G, Sarwar UN, Hu Z, Enama ME, Bailer RT, Koup RA, Schwartz RM, Akahata W, Nabel GJ, Mascola JR, Pierson TC, Graham BS, Ledgerwood JE; VRC 311 Study Team. Safety and tolerability of chikungunya virus-like particle vaccine in healthy adults: a phase 1 dose-escalation trial. Lancet. 2014 Dec 6;384(9959):2046-52. doi: 10.1016/S0140-6736(14)61185-5. Epub 2014 Aug 14. PMID 25132507
- [Background] Weaver SC, Lecuit M. Chikungunya Virus Infections. N Engl J Med. 2015 Jul 2;373(1):94-5. doi: 10.1056/NEJMc1505501. No abstract available. PMID 26132956
- [Background] Powers AM, Logue CH. Changing patterns of chikungunya virus: re-emergence of a zoonotic arbovirus. J Gen Virol. 2007 Sep;88(Pt 9):2363-2377. doi: 10.1099/vir.0.82858-0. No abstract available. PMID 17698645
- [Result] Chen GL, Coates EE, Plummer SH, Carter CA, Berkowitz N, Conan-Cibotti M, Cox JH, Beck A, O'Callahan M, Andrews C, Gordon IJ, Larkin B, Lampley R, Kaltovich F, Gall J, Carlton K, Mendy J, Haney D, May J, Bray A, Bailer RT, Dowd KA, Brockett B, Gordon D, Koup RA, Schwartz R, Mascola JR, Graham BS, Pierson TC, Donastorg Y, Rosario N, Pape JW, Hoen B, Cabie A, Diaz C, Ledgerwood JE; VRC 704 Study Team. Effect of a Chikungunya Virus-Like Particle Vaccine on Safety and Tolerability Outcomes: A Randomized Clinical Trial. JAMA. 2020 Apr 14;323(14):1369-1377. doi: 10.1001/jama.2020.2477. PMID 32286643
- [Derived] McCarty JM, Bedell L, Mendy J, Coates EE, Chen GL, Ledgerwood JE, Tredo SR, Warfield KL, Richardson JS. Chikungunya virus virus-like particle vaccine is well tolerated and immunogenic in chikungunya seropositive individuals. Vaccine. 2023 Oct 6;41(42):6146-6149. doi: 10.1016/j.vaccine.2023.08.086. Epub 2023 Sep 9. PMID 37690874

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Started | 201 | 199
Received 1st Injection | 197 | 199
Received 2nd Injection | 192 | 192
Completed | 180 | 183
Not Completed | 21 | 16
Not completed — Enrolled, but did not receive product | 4 | 0
Not completed — Lost to Follow-up | 9 | 6
Not completed — Moved from area | 2 | 3
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Physician Decision | 1 | 3
Not completed — Illness/Injury unrelated to product | 0 | 1

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP) | Total
Number analyzed (Participants) | 201 | 199 | 400
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 16 | 9 | 25
  21-30 years | 66 | 75 | 141
  31-40 years | 53 | 51 | 104
  41-50 years | 40 | 34 | 74
  51-60 years | 26 | 30 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 103 | 199
  Male | 105 | 96 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 137 | 138 | 275
  Not Hispanic or Latino | 64 | 61 | 125
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  North, South or Central American Native | 144 | 143 | 287
  Asian | 0 | 1 | 1
  Black or African American | 3 | 6 | 9
  White | 20 | 14 | 34
  More than one race | 21 | 20 | 41
  Unknown or Not Reported | 13 | 15 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  Haiti | 32 | 30 | 62
  Puerto Rico | 85 | 87 | 172
  Guadeloupe | 16 | 14 | 30
  Dominican Republic | 53 | 53 | 106
  Martinique | 15 | 15 | 30
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  under 18.5 kg/m^2 | 5 | 5 | 10
  18.5-24.9 kg/m^2 | 94 | 93 | 187
  25.0-29.9 kg/m^2 | 56 | 57 | 113
  30.0 kg/m^2 or over | 45 | 44 | 89
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Any Injection
Description: Subjects recorded the occurrence of solicited symptoms on a memory aid for 7 days after any injection and reviewed the memory aid with clinic staff at a follow up visit. Subjects are counted once for each symptom at the worst severity if they indicated experiencing the symptom at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of subjects reporting any local symptom at the worst severity. Solicited reactogenicity was recorded without an attribution assessment. Grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after any injection
Population: Population included all enrolled subjects who received at least one injection and provided safety data (via diary card and/or laboratory results) following the injection. Four subjects in Group 1 did not receive product and one subject in Group 2 did not provide a diary card following the first injection and were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Number analyzed (Participants) | 197 | 198
Participants
  Pain/Tenderness: None | 136 | 161
  Pain/Tenderness: Mild | 58 | 37
  Pain/Tenderness: Moderate | 3 | 0
  Pain/Tenderness: Severe | 0 | 0
  Swelling: None | 192 | 197
  Swelling: Mild | 2 | 0
  Swelling: Moderate | 3 | 1
  Swelling: Severe | 0 | 0
  Redness: None | 196 | 198
  Redness: Mild | 1 | 0
  Redness: Moderate | 0 | 0
  Redness: Severe | 0 | 0
  Any Local Symptom: None | 133 | 161
  Any Local Symptom: Mild | 58 | 36
  Any Local Symptom: Moderate | 6 | 1
  Any Local Symptom: Severe | 0 | 0

2. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Any Injection
Description: Subjects recorded the occurrence of solicited symptoms on a memory aid for 7 days after any injection and reviewed the memory aid with clinic staff at a follow up visit. Subjects are counted once for each symptom at the worst severity if they indicated experiencing the symptom at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of subjects reporting any systemic symptom at the worst severity. Solicited reactogenicity was recorded without an attribution assessment. Grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after any injection
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Number analyzed (Participants) | 197 | 198
Participants
  Malaise: None | 144 | 150
  Malaise: Mild | 46 | 41
  Malaise: Moderate | 7 | 7
  Malaise: Severe | 0 | 0
  Myalgia: None | 151 | 162
  Myalgia: Mild | 41 | 34
  Myalgia: Moderate | 5 | 2
  Myalgia: Severe | 0 | 0
  Headache: None | 143 | 140
  Headache: Mild | 42 | 47
  Headache: Moderate | 11 | 11
  Headache: Severe | 1 | 0
  Chills: None | 180 | 186
  Chills: Mild | 13 | 10
  Chills: Moderate | 4 | 2
  Chills: Severe | 0 | 0
  Nausea: None | 186 | 182
  Nausea: Mild | 8 | 12
  Nausea: Moderate | 3 | 4
  Nausea: Severe | 0 | 0
  Joint Pain: None | 173 | 184
  Joint Pain: Mild | 20 | 12
  Joint Pain: Moderate | 4 | 2
  Joint Pain: Severe | 0 | 0
  Temperature: None | 188 | 193
  Temperature: Mild | 7 | 2
  Temperature: Moderate | 2 | 2
  Temperature: Severe | 0 | 1
  Any Systemic Symptom: None | 110 | 113
  Any Systemic Symptom: Mild | 65 | 68
  Any Systemic Symptom: Moderate | 21 | 16
  Any Systemic Symptom: Severe | 1 | 1

3. Primary Outcome: Number of Subjects With an Abnormal Laboratory Result
Description: Safety laboratory parameters included hematology (hemoglobin, hematocrit, platelets, red blood cell (RBC), white blood cell (WBC), neutrophil, monocyte, lymphocyte, basophil and eosinophil counts, mean corpuscular volume (MCV)) and chemistry (ALT). Complete blood count, differential, platelet and ALT results were collected at screening (≤ 56 days before enrollment), Day 0 prior to study product administration (baseline), and Days 28 and 56.
Time Frame: 4 weeks after last injection
Population: Population included all enrolled subjects who had laboratory results available at any study visit post baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Number analyzed (Participants) | 194 | 197
Participants
  ALT | 7 | 4
  WBC | 21 | 18
  Hemoglobin | 50 | 70
  Platelets | 6 | 4
  Neutrophils | 32 | 30
  Lymphocytes | 7 | 4
  Eosinophils | 10 | 5
  RBC | 28 | 21
  Hematocrit | 39 | 45
  MCV | 28 | 23
  Monocytes | 5 | 6
  Basophils | 3 | 1

4. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs were reported from receipt of first study injection through 4 weeks after the last study injection administered. After the indicated time period through the last expected study visit at 72 weeks, only new chronic medical conditions and SAEs (reported as a separate outcome and in the AE module) were collected as unsolicited AEs. A subject with multiple experiences of the same event is counted once using the event of worst severity. The number reported for "Any AE" is the number of subjects reporting at least one or more AEs.
Time Frame: Through study completion, an average of 72 weeks after first injection
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Number analyzed (Participants) | 197 | 198
Participants
  Any AE | 104 | 111
  Blood and lymphatic system disorders | 45 | 46
  Cardiac disorders | 7 | 14
  Endocrine disorders | 1 | 0
  Eye disorders | 2 | 0
  Gastrointestinal disorders | 11 | 11
  General disorders & administration site conditions | 2 | 4
  Infections and infestations | 33 | 39
  Injury, poisoning & procedural complications | 6 | 4
  Investigations | 5 | 2
  Metabolism and nutrition disorders | 0 | 1
  Musculoskeletal and connective tissue disorders | 5 | 4
  Neoplasms benign, malignant and unspecified | 0 | 1
  Nervous system disorders | 3 | 4
  Pregnancy, puerperium & perinatal conditions | 1 | 0
  Psychiatric disorders | 1 | 0
  Renal and urinary disorders | 0 | 2
  Reproductive system and breast disorders | 0 | 2
  Respiratory, thoracic and mediastinal disorders | 9 | 4
  Skin and subcutaneous tissue disorders | 3 | 9
  Surgical and medical procedures | 1 | 1
  Vascular disorders | 15 | 13

5. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs were reported from receipt of first study injection through the last expected study visit at 72 weeks. Grading (Mild, Moderate, Severe, Life-threatening, and Death) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007). The relationship between a SAE and the study product was assessed by the investigator on the basis of his or her clinical judgment and the definitions outlined in the protocol. A subject with multiple SAEs is counted only once.
Time Frame: Through study completion, an average of 72 weeks after first injection
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Number analyzed (Participants) | 197 | 198
Participants
  Related to study product | 0 | 0
  Unrelated to study product | 4 | 11

6. Primary Outcome: Number of Subjects With Confirmed Chikungunya Virus (CHIKV) Infection Events
Description: Confirmed Chikungunya infections by positive polymerase chain reaction (PCR) results reported from receipt of first study injection through the last expected study visit at 72 weeks.
Time Frame: Through study completion, an average of 72 weeks after first injection
Population: Population included all enrolled subjects who received at least one injection. Four subjects in Group 1 did not receive product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Number analyzed (Participants) | 197 | 199
Participants | 1 | 0

7. Secondary Outcome: Chikungunya Antigen-specific Neutralizing Antibody Geometric Mean Titer (GMT) - Per Protocol Population
Description: Antibody responses as measured by neutralization antibody (NAb) assay 4 weeks after last study injection.
Time Frame: Week 8
Population: Subjects who received 2 injections within window as assigned by the randomization schedule and didn't experience any other major protocol deviations prior to Week 8 visit, including those that were CHIKV-infected prior to receipt of 2nd injection who didn't experience deviations prior to infection. None were CHIKV-infected prior to 2nd injection.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Number analyzed (Participants) | 182 | 181
titer | 2088.2 [1765.2 to 2474.1] | 41.1 [30.3 to 55.8]

8. Secondary Outcome: Chikungunya Antigen-specific Neutralizing Antibody Geometric Mean Titer (GMT) - Intent-to-Treat Population
Description: Antibody responses as measured by neutralization antibody (NAb) assay 4 weeks after last study injection.
Time Frame: Week 8
Population: Intent-to-Treat (ITT) population included all enrolled subjects, analyzed according to the randomized vaccine, with immunogenicity data.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Number analyzed (Participants) | 193 | 193
titer | 1995.7 [1673.9 to 2379.3] | 42.6 [31.6 to 57.5]

9. Secondary Outcome: Chikungunya Antigen-specific Neutralizing Antibody Geometric Mean Titer (GMT) - Modified Intent-to-Treat
Description: Antibody responses as measured by neutralization antibody (NAb) assay 4 weeks after last study injection.
Time Frame: 4 weeks after last study injection
Population: Modified Intent-to-Treat (mITT) population included all enrolled subjects who received at least one injection with non-missing immunogenicity data at their Week 8 visit, without exclusions for protocol deviations or censoring for CHIKV infection
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
Number analyzed (Participants) | 192 | 192
titer | 2004.5 [1680.1 to 2391.5] | 42.8 [31.7 to 57.9]

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after any injection. Unsolicited AEs were reported from receipt of the first injection through 4 weeks after the last study injection administered. Following the time period defined for AEs through the last expected study visit at 72 weeks, only new chronic medical conditions were collected as unsolicited AEs. Serious AEs (SAEs) were reported from receipt of the first injection through the last expected study visit at 72 weeks.
Description: Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment are reported by subjects who received at least one injection and provided safety data following the injection, and represent the number and percentage of subjects reporting the event. A subject with multiple experiences of the same event is counted once using the event of worst severity. A subject with multiple SAEs is counted only once.
Arm/Group | Group 1: VRC-CHKVLP059-00-VP 20 mcg | Group 2: Placebo (VRC-PBSPLA043-00-VP)
All-Cause Mortality (participants affected / at risk) | 0/197 | 0/198
Serious Adverse Events (participants affected / at risk) | 4/197 | 11/198
Other Adverse Events (participants affected / at risk) | 123/197 | 128/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: VRC-CHKVLP059-00-VP 20 mcg (N=197) | Group 2: Placebo (VRC-PBSPLA043-00-VP) (N=198)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Appendicectomy (Surgical and medical procedures) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Acute hepatitis B (Infections and infestations) | 0 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1
Near drowning (Injury, poisoning and procedural complications) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: VRC-CHKVLP059-00-VP 20 mcg (N=197) | Group 2: Placebo (VRC-PBSPLA043-00-VP) (N=198)
Anaemia (Blood and lymphatic system disorders) | 20 | 29
Neutropenia (Blood and lymphatic system disorders) | 10 | 10
Bradycardia (Cardiac disorders) | 5 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 13
Administration Site Pain/Tenderness (General disorders) | 61 | 37
Malaise (General disorders) | 53 | 48
Myalgia (Musculoskeletal and connective tissue disorders) | 46 | 36
Headache (Nervous system disorders) | 54 | 58
Chills (General disorders) | 17 | 12
Nausea (Gastrointestinal disorders) | 11 | 16
Joint Pain (Musculoskeletal and connective tissue disorders) | 24 | 14

LIMITATIONS AND CAVEATS:
Exploratory immunogenicity analyses (to evaluate humoral and cellular responses to VRC-CHKVLP059-00-VP at additional time points by antibody assays that include antigen-specific ELISA and neutralization assay) were not completed and are not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT02562482/Prot_SAP_ICF_001.pdf